CLINICAL TRIAL: NCT02250300
Title: MLN9708 for the Prophylaxis of Chronic Graft-versus-host Disease in Patient Undergoing Allogeneic Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mehdi Hamadani (Other)
Responsible Party: Sponsor-Investigator, Mehdi Hamadani, Associate Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00022660
Record Dates: First submitted 2014-08-07; First posted 2014-09-26 (Estimated); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-01

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Stem cell transplantation; Hematopoietic transplantation; Hematopoietic stem cell
MeSH Terms: interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MLN9708 Phase II matched sibling (Experimental): Phase II Patients will be enrolled in two independent cohorts of matched sibling and matched unrelated donor transplants. Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 starting on day +60 to +90 post allogeneic HCT.
  Interventions: Drug: MLN9708 (4.0 mg)
- MLN9708 Phase II matched unrelated (Experimental): Phase II Patients will be enrolled in two independent cohorts of matched sibling and matched unrelated donor transplants. Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 starting on day +60 to +90 post allogeneic HCT.
  Interventions: Drug: MLN9708 (4.0 mg)
- MLN9708 Phase I (2.3 mg) (Experimental): Phase I Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 orally based on a dose escalation schema.
  Interventions: Drug: MLN9708 (2.3 mg)
- MLN9708 Phase I (3.0 mg) (Experimental): Phase I Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 orally based on a dose escalation schema.
  Interventions: Drug: MLN9708 (3.0 mg)
- MLN9708 Phase I (4.0 mg) (Experimental): Phase I Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 orally based on a dose escalation schema.
  Interventions: Drug: MLN9708 (4.0 mg)

INTERVENTIONS:
Drug: MLN9708 (2.3 mg) — 2.3 mg
  Other Names: Ixazomib
  Arms: MLN9708 Phase I (2.3 mg)
Drug: MLN9708 (4.0 mg) — 4.0 mg
  Other Names: Ixazomib
  Arms: MLN9708 Phase I (4.0 mg); MLN9708 Phase II matched sibling; MLN9708 Phase II matched unrelated
Drug: MLN9708 (3.0 mg) — 3.0 mg
  Other Names: Ixazomib
  Arms: MLN9708 Phase I (3.0 mg)

SUMMARY:
This is a phase I/II study of MLN9708 for the prophylaxis of chronic graft-versus-host-disease (GVHD) in patients undergoing allogeneic hematopoietic stem cell transplantation (HSCT).

During the phase I portion, patients undergoing both sibling and unrelated donor transplantation will be enrolled on the same arm to determine the dose-limiting toxicity (DLT) and maximum-tolerated dose (MTD).

During the phase II portion of the trial, patients will be enrolled into two separate and independent cohorts: a) Matched sibling transplants and b) Unrelated donors transplants. Both cohorts will be enrolled and analyzed separately.

DETAILED DESCRIPTION:
* For potential candidates for this trial, the recommended acute GVHD prophylaxis is a tacrolimus, methotrexate and atorvastatin combination. However, any acute GVHD prophylaxis regimen at the discretion of treating physician (not involving in vivo or ex vivo T-cell depletion, cluster of differentiation 34 (CD34) + cell selection, or post-HCT cyclophosphamide) will be permitted.
* During the phase I portion for chronic GVHD prophylaxis, four doses of MLN9708 will be administered orally (to patients undergoing either matched sibling or unrelated donor transplantation) on days 1, 8, 15 and 22, starting on day +60 to +74 post allogeneic HCT.

If zero of three patients experienced DLT at dose level 2, then it would be considered a MTD. If two or more patients experienced a DLT, dose escalation would halt and the dose level would be expanded to six patients to determine the MTD. If the dose level below already has six patients, enrolled, then it will be considered the MTD. If two or more patients experience DLT on first dose level (i.e., dose level 1), then, patients will be enrolled on dose level -1. No intrapatient dose escalation will be permitted.

* MTD is defined at maximum dose level with fewer than two of six patients experiencing DLT.
* The phase II portion will utilize the MTD for MLN9708, determined from phase I portion of the study. In phase II, patients will be enrolled in two independent cohorts of matched sibling and matched unrelated donor transplants.
* During the phase II portion, for chronic GVHD prophylaxis, four doses of MLN9708 will be administered orally on days 1, 8, 15 and 22, starting on day +60 to +90 post allogeneic HCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of a hematological malignancy or bone marrow failure syndrome undergoing (or status post) a peripheral blood allogeneic HCT.
2. Patients aged ≥18 are eligible.
3. All patients must have received or plan to receive an allograft from a suitable human leukocyte antigens (HLA) -matched sibling or unrelated donor according to transplant center's guidelines (for selection of appropriate donor).
4. Voluntary written consent must be given before patient registration and performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
5. Bilirubin ≤ 2 x the upper limit of normal (ULN). For patients with Gilbert's syndrome or suspected mild veno-occlusive disease, bilirubin ≤ 3 x ULN is permitted.
6. Creatinine clearance of ≥ 30 mL/min calculated by Cockcroft-Gault equation.
7. Karnofsky performance status > 60.
8. A negative pregnancy test will be required for all women of child bearing potential. Females of child bearing potential should agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug and must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.). Breast feeding is not permitted.
9. Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following: practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
10. No evidence of uncontrolled bacterial, viral or fungal infections at the time of enrollment.
11. No known active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.

Exclusion Criteria:

1. Patients with active ≥ grade 3 peripheral neuropathy or grade 2 with pain on clinical examination during the screening period will be excluded.
2. Patients with history of allergy and/or intolerance to MLN9708 are not eligible.
3. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing is not permitted.
4. Patients receiving (or status post) a cord blood or a haplo-identical allograft will not be eligible.
5. Patients undergoing (or status post) a T-cell depleted allogeneic transplantation will not be eligible.
6. Patients receiving (or status post) conditioning regimens containing antithymocyte globulin, and/or campath, one receiving post-HCT planned cyclophosphamide will not be eligible.
7. Method of stem-cell collection from the donor will be at the discretion of the treating physician. Although it is anticipated that majority of patients will receive allograft mobilized with Granulocyte- colony stimulating factor (CSF) alone; however donors receiving allografts mobilized with experimental agents (e.g. plerixafor) will remain eligible for the study.
8. Patients experiencing disease relapse (for those in complete remission at the time of HCT) or progression (for those in partial remission, stable or refractory disease at the time of HCT) will be excluded.
9. Donor lymphocyte infusions between day zero of HCT and first dose of MLN9708 are not permitted.
10. Rituximab (or other B-cell depleting monoclonal antibodies) or bortezomib administration between day zero of HCT and before the first day of MLN9708 is not permitted.
11. Patients with steroid refractory (defined as no improvement of symptoms after 7 days of systemic corticosteroids at a dose of ≥1mg/kg/day) grade II-IV acute GVHD, that is active at the time of enrollment will be excluded.
12. Patients with grade III-IV acute GVHD (even if it is not meeting criteria for steroid refractory acute GVHD), that is active at the time of enrollment will be excluded. Patients with controlled grade I-II acute GVHD can be enrolled after discussing with study PI. Topical or systemic corticosteroids therapy, as per standard of care for such grade I-II acute GVHD patients is permitted.
13. Patients with active chronic GVHD (although unlikely before day +100) will be excluded.
14. No major surgery within 14 days before enrollment.
15. No radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708.
16. No evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months. Cardiac enzyme elevations for reasons other than document myocardial infarction is not an exclusion.
17. No systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450, family 3, subfamily A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
18. No serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
19. No participation in other clinical trials, including those with other investigational agents within 21days of the start of this trial and throughout the duration of this trial. However co-enrollment on trials evaluating conditioning regimens, institutional protocols evaluating atorvastatin for acute GVHD prophylaxis, and stem cell collection protocols in transplant donors will be permitted. In addition patients randomized to standard-of-care (non experimental) arms of available phase II/III trials will be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Hamadani, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chhabra S, Visotcky A, Pasquini MC, Zhu F, Tang X, Zhang MJ, Thompson R, Abedin S, D'Souza A, Dhakal B, Drobyski WR, Fenske TS, Jerkins JH, Douglas Rizzo J, Runaas L, Saber W, Shah NN, Shaw BE, Horowitz MM, Hari PN, Hamadani M. Ixazomib for Chronic Graft-versus-Host Disease Prophylaxis following Allogeneic Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2020 Oct;26(10):1876-1885. doi: 10.1016/j.bbmt.2020.07.005. Epub 2020 Jul 9. PMID 32653622

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven of the 68 subjects consenting to participate were determined to be ineligible to participate in the study. The remaining 57 total subjects are detailed below. The initial dose of MLN9708 in the escalation phase was 3.0mg. Due to no DLTs experienced in this group, no subjects were enrolled to the lower 2.3mg cohort.
Groups:
- MLN9708 Phase I (3.0 mg): Phase I Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 orally based on a dose escalation schema.
  MLN9708 (3.0 mg)
- MLN9708 Phase I (4.0 mg): Phase I Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 orally based on a dose escalation schema.
  MLN9708 (4.0 mg)
Period: Dose Escalation 3.0 mg Phase
Arm/Group | MLN9708 Phase II Matched Sibling | MLN9708 Phase II Matched Unrelated | MLN9708 Phase I (3.0 mg) | MLN9708 Phase I (4.0 mg)
Started | 0 | 0 | 3 | 0
Completed | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Escalation 4.0 mg Phase
Arm/Group | MLN9708 Phase II Matched Sibling | MLN9708 Phase II Matched Unrelated | MLN9708 Phase I (3.0 mg) | MLN9708 Phase I (4.0 mg)
Started | 0 | 0 | 0 (This cohort was involved only in the 3.0 mg dose escalation phase and were not involved in subsequent phases of the study.) | 3 (This cohort was involved only in the 4.0 mg dose escalation phase and were not involved in prior or subsequent phases of the study.)
Completed | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Expansion Phase
Arm/Group | MLN9708 Phase II Matched Sibling | MLN9708 Phase II Matched Unrelated | MLN9708 Phase I (3.0 mg) | MLN9708 Phase I (4.0 mg)
Started | 25 (This expansion cohort involved a new group of subjects using the 4.0 mg dose.) | 26 (This expansion cohort involved a new group of subjects using the 4.0 mg dose.) | 0 | 0 (This cohort was involved only in the 4.0 mg dose escalation phase and was not involved in expansion phase of the study.)
Completed | 19 | 19 | 0 | 0
Not Completed | 6 | 7 | 0 | 0
Not completed — Death | 6 | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MLN9708 Phase II Matched Sibling: Phase II Patients will be enrolled in two independent cohorts of matched sibling and matched unrelated donor transplants. Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 starting on day +60 to +90 post allogeneic hematopoietic cell transplant (HCT).
  MLN9708 (4.0 mg): 4.0 mg
- Total: Total of all reporting groups
Arm/Group | MLN9708 Phase II Matched Sibling | MLN9708 Phase II Matched Unrelated | MLN9708 Phase I (3.0 mg) | MLN9708 Phase I (4.0 mg) | Total
Number analyzed (Participants) | 25 | 26 | 3 | 3 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 1 | 1 | 44
  >=65 years | 3 | 6 | 2 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.3) | 53.5 (12.9) | 65.3 (0.9) | 65.0 (8.0) | 53.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 2 | 1 | 17
  Male | 18 | 19 | 1 | 2 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 26 | 3 | 3 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 24 | 26 | 3 | 3 | 56
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 3 | 3 | 57

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose of MLN9708.
Description: Maximum-tolerated dose of ixazomib (MLN9708) will be determined from the incidence of dose limiting toxicities at each dosage. Results for both escalation phase cohorts (3.0 mg and 4.0 mg) were used to determine the maximum tolerated dose.
Time Frame: 4 weeks
Population: Only the subjects in the Phase I dose escalation study are included in this outcome measure.
Measure: Number; unit: millligram
Groups:
- Maximum Tolerated Dose of Study Drug: This measure is the maximum dosage of study drug based on the count of Drug Limiting Toxicities (DLT). The number of DLT for each dosage are listed in the results of Outcome Measure #3.
Arm/Group | Maximum Tolerated Dose of Study Drug
Number analyzed (Participants) | 6
millligram | 4

2. Primary Outcome: Cumulative Incidence of Chronic Graft-versus-host Disease.
Description: The number of participants who have graft-versus-host disease. The two expansion phase cohorts (3.0 mg and 4.0 mg) were not included in this analysis.
Time Frame: 1 year
Population: The Phase 1 dose escalation cohort is not included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MLN9708 Phase II Matched Sibling | MLN9708 Phase II Matched Unrelated
Number analyzed (Participants) | 25 | 26
Participants | 9 | 10

3. Primary Outcome: Number of Participants Experiencing Dose-limiting Toxicity of MLN9708
Description: A 3+3 design will be employed. At each dose, three patients will be initially evaluated. If no dose limiting toxicities are observed, the MLN9708 dose will be increased; if one dose limiting toxicity is observed, three additional patients will be treated at that dose. A dose at which two DLTs are observed in three or six patients are judged to be too toxic, the lower dose will be defined as the maximally tolerated dose (MTD).
Time Frame: 4 weeks
Population: Based on the escalation schema and lack of dose limiting toxicities, the 2.3mg dosage cohort was not required.
Measure: Number; unit: dose limiting toxicity
Arm/Group | MLN9708 Phase I (3.0 mg) | MLN9708 Phase I (4.0 mg)
Number analyzed (Participants) | 3 | 3
dose limiting toxicity | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for the Phase 1 cohort for four weeks. Adverse events for the remaining cohorts were collected up to one year.
Description: One subject in the Phase 1 cohort expired after the 4 week dose escalation phase but prior to the end of study data collection.
Groups:
- MLN9708 Phase I (3.0mg): Phase I Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 orally based on a dose escalation schema.
  MLN9708 (3.0 mg)
- MLN9708 Phase I (4.0mg): Phase I Four doses of MLN9708 will be administered on days 1, 8, 15, & 22 orally based on a dose escalation schema.
  MLN9708 (4.0 mg)
Arm/Group | MLN9708 Phase II Matched Sibling | MLN9708 Phase II Matched Unrelated | MLN9708 Phase I (3.0mg) | MLN9708 Phase I (4.0mg)
All-Cause Mortality (participants affected / at risk) | 6/25 | 7/26 | 1/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 6/25 | 17/26 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 25/25 | 26/26 | 2/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLN9708 Phase II Matched Sibling (N=25) | MLN9708 Phase II Matched Unrelated (N=26) | MLN9708 Phase I (3.0mg) (N=3) | MLN9708 Phase I (4.0mg) (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Chemotherapy induced cardiomyopathy with left ventricular systolic dysfunction
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Vancomycin resistant enterococcus
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLN9708 Phase II Matched Sibling (N=25) | MLN9708 Phase II Matched Unrelated (N=26) | MLN9708 Phase I (3.0mg) (N=3) | MLN9708 Phase I (4.0mg) (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 8 (8) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Investigations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 8 (8) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 11 (11) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (7) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter-related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT02250300/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT02250300/ICF_001.pdf